CLINICAL TRIAL: NCT00739557
Title: A Pilot Study to Evaluate the Systemic Inflammatory Response of Thoracoabdominal Aortic Aneurysm Repair.
Status: Withdrawn | Type: Observational
Why Stopped: Investigator left the institution, another PI has not been named.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Other Study IDs: 07-0257
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Aortic Aneurysm, Thoracic; Systemic Inflammatory Response Syndrome
Keywords: elective TAAA repair
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and saliva samples will be obtained for the purposes of this study and will be maintained until complete analysis of the samples for all patients is complete.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to look at the systemic inflammatory response caused when patients undergo thoracoabdominal aortic aneurysm repair (TAAA). In addition, this study will look at how the inflammatory response affects the post operative healing process and post operative complications.

DETAILED DESCRIPTION:
Patients will be invited to participate in this study prior to the TAAA repair procedure. Prior to the surgery, baseline blood and saliva samples will be collected. Following the surgery, blood and saliva samples will be collected for 48 hours. In addition, hemodynamic data (i.e. vital signs) will be collected for the first 48 hours. The patient data will be reviewed for the first 30 days for morbidity and mortality assessment.

ELIGIBILITY:
Inclusion Criteria:

* Elective TAAA repair

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients entering the hospital for elective TAAA repair
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
to evaluate the effects of TAAAA repair on pro-inflammatory mediators and the anti-inflammatory mediators IL-1 receptor antagonist and IL-10. | 30 days

SECONDARY OUTCOMES:
To characterize the inflammatory response after TAAA repair and delineate any association to post-operative morbidity | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth S Helmer, MD, Principal Investigator — Univ. of Texas Health Science Center at Houston